CLINICAL TRIAL: NCT04849143
Title: The Effectiveness of Stingless Bee Honey (Kelulut Honey) Dressing Versus Conventional Gel Dressing for Wound Bed Preparation in Diabetic Patients With Cavity Wounds: A Randomised Controlled Trial
Brief Title: The Effectiveness of Stingless Bee Honey (Kelulut Honey) Versus Gel in Diabetic Wound Bed Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohamad Aizat Bin Rosli, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/21020186
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus; Wound Heal; Diabetes; Honey
MeSH Terms: conditions — Diabetes Mellitus | interventions — aloe vera gel extract hydrogel dressing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey dressing group (Experimental): A thin layer of honey will be applied to the wounds
  Interventions: Other: Stingless bee honey ( Kelulut honey)
- Gel dressing group (Active Comparator): A thin layer of gel will be applied to the wounds
  Interventions: Other: Gel dressing

INTERVENTIONS:
Other: Stingless bee honey ( Kelulut honey) — The honey will be acquired from Brainey Sdn Bhd, a company that provides stingless bee honey certified with Good Manufacturing Practice (GMP), ISO 22000, and Halal.
  As the honey used is not medical-grade honey, sterilization with 25kGy gamma-ray irradiation will be done for safety purposes to eradicate any potential life-threatening infection such as spores from Clostridium botulinum.
  Arms: Honey dressing group
Other: Gel dressing — Smith-Nephew's Intrasite gel
  Arms: Gel dressing group

SUMMARY:
There has been no study yet on the effect of stingless bee honey (Kelulut honey) produced by Melipolini sp. in diabetic wound healing in Malaysia. Kelulut honey, apart from possessing similar pro-healing properties with other honey, is also found to have a better antioxidant capacity, anti-inflammatory, and free radical scavenging activity than Tualang honey. These effects are due to the much higher content of phenolic and flavonoid substances in Kelulut honey, the key bioactive factors promoting wound healing and preventing oxidative stress-related injury. Australian researchers have also recently discovered a novel source of the rare disaccharide trehalose in stingless bee's honey, which is highly anti-diabetic and antioxidating. This study aims to investigate the efficacy of honey against gel dressing for wound bed preparation among diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Aged between 18-70 years old
* Patient with full thickness cavity wound
* Controlled diabetes mellitus (defined as: fasting blood glucose (FBG) < 10 mmol/L upon selection)

Exclusion Criteria:

* Severely contaminated wound/infected
* Patient with history of allergy to honey or stingless bee product
* Patients who are immunocompromised or on chronic steroid use ( defined as use of steroid for more than 2 weeks)
* Pregnancy
* End stage renal failure (ESRF) patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Size of granulation tissue | 30 days
  This will be calculated based on the surface area of granulation tissue traced and marked on the Opsite Flexigrid by indelible fine tip marker. The amount of small squares will calculated and this will represent the surface area. The change between baseline and at day 30 will be recorded as percentage.
Wound size reduction | 30 days
  This will be calculated based on the surface area of the whole wound traced and marked on the Opsite Flexigrid by indelible fine tip marker. The amount of small squares will calculated and this will represent the surface area. The change between baseline and at day 30 will be recorded as percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Aizat Rosli, MB ChB, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No